CLINICAL TRIAL: NCT07087184
Title: Gauging Outcomes of Total Milk Ingestion on Lipid and gControl
Acronym: GOT MILC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 25-44169
Record Dates: First submitted 2025-07-18; First posted 2025-07-25 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Heart Diseases; Cardiovascular Disease
Keywords: Cardiovascular Disease; Milk Fat; Milk; Dairy Products; Insulin Resistance; Hyperlipidemia
MeSH Terms: conditions — Heart Diseases; Cardiovascular Diseases; Insulin Resistance; Hyperlipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole Milk-Skim Milk (Experimental): Participants randomized to the whole milk-skim milk treatment sequence will be instructed to limit their liquid milk consumption to only whole milk during the first two months of the study (Month 1-2), followed by only non-fat milk during the final two months of the study (Month 3-4). Using an N-of-1 strategy delivered by the National Institutes of Health (NIH)-funded, University of California, San Francisco (UCSF)-run Eureka platform utilizing a mobile smartphone-based application, subjects will be instructed weekly via app and text-based messaging on the type of liquid milk (whole or non-fat) to consume.
  Interventions: Behavioral: Whole Milk-Skim Milk
- Skim Milk-Whole Milk (Experimental): Participants randomized to the skim milk-whole milk treatment sequence will be instructed to limit their liquid milk consumption to only non-fat milk during the first two months of the study (Month 1-2), followed by only whole-fat milk during the final two months of the study (Month 3-4). Using an N-of-1 strategy delivered by the National Institutes of Health (NIH)-funded, University of California, San Francisco (UCSF)-run Eureka platform utilizing a mobile smartphone-based application, subjects will be instructed weekly via app and text-based messaging on the type of liquid milk (whole or non-fat) to consume.
  Interventions: Behavioral: Skim Milk-Whole Milk

INTERVENTIONS:
Behavioral: Whole Milk-Skim Milk — If randomized to the whole milk-skim milk treatment sequence, participants will be instructed to restrict their liquid milk consumption to only whole milk for the first 2 months and to only skim milk for the last 2 months of the enrollment period. Participants will receive weekly app and text-based message reminders of their randomization assignments.
  Arms: Whole Milk-Skim Milk
Behavioral: Skim Milk-Whole Milk — If randomized to the skim milk-whole milk treatment sequence, participants will be instructed to restrict their liquid milk consumption to only skim milk for the first 2 months and to only whole milk for the last 2 months of the enrollment period. Participants will receive weekly app and text-based message reminders of their randomization assignments.
  Arms: Skim Milk-Whole Milk

SUMMARY:
Atherosclerotic cardiovascular disease remains the leading cause of death for adults in the United States. The cardiovascular impact of milk consumption remains a matter of long-standing scientific debate. Current guidelines for Americans recommend three daily servings of fat-free or low-fat (1%) dairy over full-fat options due to concerns that saturated fat may increase cardiovascular risk. Yet, the literature does not consistently support non-fat dairy as superior to high-fat dairy for reducing cardiometabolic risk. Identifying the comparative health benefits of non-fat versus high-fat dairy milk would be immediately applicable to patients who seek cardiovascular care. In this randomized, case-crossover trial, the investigators seek to efficiently assess the association between high-fat versus non-fat dairy milk consumption and insulin resistance. Utilizing the Eureka Platform, participants will be randomized to limit their liquid milk consumption to whole milk followed by skim milk (or vice versa), measuring the effect of milk fat content on glycemic index and lipid profile.

DETAILED DESCRIPTION:
The study is designed as an N of 1 randomized trial, where each participant will be randomized to consume high-fat versus non-fat dairy milk then crossover to the alternate condition over two consecutive two-month periods. After two and four months, participants will have lab tests performed, including hemoglobin A1c (HbA1c) and fasting lipids. Throughout the study, participants will be instructed to continuously wear a wrist-worn fitness tracker, use a Bluetooth-enabled scale and blood pressure monitor to trend weight and blood pressure weekly, and utilize the Eureka mobile application for self-monitoring of dairy milk consumption, diet, lifestyle, and physical activity. Aside from study-related dairy milk instructions, all other aspects of diet will remain constant throughout study participation. The study seeks to elucidate the relationship between dairy milk consumption and overall health. A total of 100 participants will be enrolled for participation in this clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Are age ≥18 years
* Have a smartphone
* Are able to use the Eureka mobile application
* Consume, on average, at least one cup of dairy milk daily, at least 5 days per week

Exclusion Criteria:

* Non-English speaker
* Are lactose intolerant
* History of myocardial infarction
* History of type I or type II diabetes
* Familial hypercholesterolemia
* Plan to change treatment for cholesterol
* Unable to read or sign to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-24 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Difference in hemoglobin A1c (HbA1c) | Measured at 2 months and 4 months after intervention initiation
  The primary outcome will be a difference in hemoglobin A1c (HbA1c) with whole-fat milk compared to skim milk during the enrollment period.

SECONDARY OUTCOMES:
Change in fasting lipid profile with whole-fat milk compared to skim milk | Measured at 2 months and 4 months after intervention initiation
  A secondary outcome will be a change in fasting lipid profile with whole-fat milk compared to skim milk during the enrollment period.
Change in blood pressure with whole-fat milk compared to skim milk | Measured weekly over the 4-month trial enrollment
  Participants will receive weekly instruction via app or text-based messaging to utilize a Bluetooth blood pressure monitor in the morning prior to taking any medication. A secondary outcome will be a change in diastolic, systolic, and mean blood pressure with whole-fat milk compared to skim milk.
Change in body weight with whole-fat milk compared to skim milk | Measured weekly over the 4-month trial enrollment
  Participants will receive weekly instruction via app or text-based messaging to utilize a Bluetooth scale in the morning prior to the first meal of the day. A secondary outcome will be a change in body weight with whole-fat milk compared to skim milk.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory M Marcus, MD, MAS, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Medical Center at Parnassus, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hoyt G, Hickey MS, Cordain L. Dissociation of the glycaemic and insulinaemic responses to whole and skimmed milk. Br J Nutr. 2005 Feb;93(2):175-7. doi: 10.1079/bjn20041304. PMID 15788109
- [Background] Drouin-Chartier JP, Cote JA, Labonte ME, Brassard D, Tessier-Grenier M, Desroches S, Couture P, Lamarche B. Comprehensive Review of the Impact of Dairy Foods and Dairy Fat on Cardiometabolic Risk. Adv Nutr. 2016 Nov 15;7(6):1041-1051. doi: 10.3945/an.115.011619. Print 2016 Nov. PMID 28140322
- [Background] Astrup A, Magkos F, Bier DM, Brenna JT, de Oliveira Otto MC, Hill JO, King JC, Mente A, Ordovas JM, Volek JS, Yusuf S, Krauss RM. Saturated Fats and Health: A Reassessment and Proposal for Food-Based Recommendations: JACC State-of-the-Art Review. J Am Coll Cardiol. 2020 Aug 18;76(7):844-857. doi: 10.1016/j.jacc.2020.05.077. Epub 2020 Jun 17. PMID 32562735
- [Background] Aune D, Norat T, Romundstad P, Vatten LJ. Dairy products and the risk of type 2 diabetes: a systematic review and dose-response meta-analysis of cohort studies. Am J Clin Nutr. 2013 Oct;98(4):1066-83. doi: 10.3945/ajcn.113.059030. Epub 2013 Aug 14. PMID 23945722
- [Background] Pereira MA, Jacobs DR Jr, Van Horn L, Slattery ML, Kartashov AI, Ludwig DS. Dairy consumption, obesity, and the insulin resistance syndrome in young adults: the CARDIA Study. JAMA. 2002 Apr 24;287(16):2081-9. doi: 10.1001/jama.287.16.2081. PMID 11966382
- [Background] Dehghan M, Mente A, Rangarajan S, Sheridan P, Mohan V, Iqbal R, Gupta R, Lear S, Wentzel-Viljoen E, Avezum A, Lopez-Jaramillo P, Mony P, Varma RP, Kumar R, Chifamba J, Alhabib KF, Mohammadifard N, Oguz A, Lanas F, Rozanska D, Bostrom KB, Yusoff K, Tsolkile LP, Dans A, Yusufali A, Orlandini A, Poirier P, Khatib R, Hu B, Wei L, Yin L, Deeraili A, Yeates K, Yusuf R, Ismail N, Mozaffarian D, Teo K, Anand SS, Yusuf S; Prospective Urban Rural Epidemiology (PURE) study investigators. Association of dairy intake with cardiovascular disease and mortality in 21 countries from five continents (PURE): a prospective cohort study. Lancet. 2018 Nov 24;392(10161):2288-2297. doi: 10.1016/S0140-6736(18)31812-9. Epub 2018 Sep 11. PMID 30217460
- [Background] Martin SS, Aday AW, Almarzooq ZI, Anderson CAM, Arora P, Avery CL, Baker-Smith CM, Barone Gibbs B, Beaton AZ, Boehme AK, Commodore-Mensah Y, Currie ME, Elkind MSV, Evenson KR, Generoso G, Heard DG, Hiremath S, Johansen MC, Kalani R, Kazi DS, Ko D, Liu J, Magnani JW, Michos ED, Mussolino ME, Navaneethan SD, Parikh NI, Perman SM, Poudel R, Rezk-Hanna M, Roth GA, Shah NS, St-Onge MP, Thacker EL, Tsao CW, Urbut SM, Van Spall HGC, Voeks JH, Wang NY, Wong ND, Wong SS, Yaffe K, Palaniappan LP; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. 2024 Heart Disease and Stroke Statistics: A Report of US and Global Data From the American Heart Association. Circulation. 2024 Feb 20;149(8):e347-e913. doi: 10.1161/CIR.0000000000001209. Epub 2024 Jan 24. PMID 38264914
- [Background] Lanou AJ, Barnard ND. Dairy and weight loss hypothesis: an evaluation of the clinical trials. Nutr Rev. 2008 May;66(5):272-9. doi: 10.1111/j.1753-4887.2008.00032.x. PMID 18454813
- [Background] Thorning TK, Raben A, Tholstrup T, Soedamah-Muthu SS, Givens I, Astrup A. Milk and dairy products: good or bad for human health? An assessment of the totality of scientific evidence. Food Nutr Res. 2016 Nov 22;60:32527. doi: 10.3402/fnr.v60.32527. eCollection 2016. PMID 27882862
- [Background] U.S. Department of Agriculture and U.S. Department of Health and Human Services. Dietary Guidelines for Americans, 2020-2025. 9th Edition. December 2020. Available at DietaryGuidelines.gov.